CLINICAL TRIAL: NCT01910623
Title: Long-Term Quality of Life in Patients With Acute Promyelocytic Leukemia: a Follow-up Observational Study of Patients Enrolled in the GIMEMA AIDA 0493 and AIDA 200
Brief Title: Long-Term Quality of Life in Patients With Acute Promyelocytic Leukemia
Acronym: QOL-APL0512
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QOL-APL0512
Record Dates: First submitted 2013-03-28; First posted 2013-07-29 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Quality of life; Health related quality of life outcomes; Long-term; Aida 0493; AIDA 2000
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Quality of Life; Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients being studied: APL patients previously enrolled in GIMEMA AIDA 0493 and AIDA 2000 studies.
  Interventions: Other: Health Related Quality of Life (HRQOL) measures

INTERVENTIONS:
Other: Health Related Quality of Life (HRQOL) measures
  Other Names: SF-36 health survey.; EORTC QOL-C30 questionnaire.; FACIT-Fatigue questionnaire.; Self-administered Comorbidity Questionnaire (SCQ).; Multidimensional Scale of Perceived Social Support (MSPSS).; MD Anderson Symptom Inventory (MDASI).

SUMMARY:
This study will focus on acute promyelocytic leukemia patients who have been diagnosed more than 5 years ago and their present quality of life.

The possible late effects of cancer treatment can include several issues and, thus, there has been an increasing interest worldwide in studying the long-term impact of these in patients' life.

DETAILED DESCRIPTION:
This study will focus on long-term survivors as defined by the America Cancer Society, that is surviving the initial diagnosis for more than 5 years. Previous research has investigated long-term Health Related Quality of Life (HRQOL) in patients with acute myeloid leukemia, however, this will be the first research conducted to investigate long-term HRQOL outcomes in patients with acute promyelocytic leukemia (APL).

The potential late effects of cancer treatment can include second malignancies or other chronic conditions affecting physical and emotional well-being. Therefore, there has been an increasing interest worldwide in evaluating the longer-term impact of cancer and its treatment. Currently large cohort of patients enjoys disease-free survival of 5 years or longer. However, a disease-free status is not synonymous with a life free of physical and psychological health related to the cancer and/or its treatment. Research shows that cancer related health concerns persist long after initial treatment and this has been shown in several cancer populations including prostate, testicular, breast cancer and lymphoma patients. Long-term cancer survivors can experience treatment-induced morbidity (e.g. cardiovascular damage due to chemotherapy or radiotherapy; infertility and second tumors), chronic disease and treatment-related symptoms, functional impairment, psychosocial problems, and practical problems.

Since the introduction of the vitamin A derivative all-trans retinoic acid (ATRA) as front-line therapy for APL, the outcome of this acute leukemia subtype has changed from the state of a most frequently fatal leukemia to the condition of a highly curable disease. The Italian cooperative group GIMEMA designed in 1993 the AIDA (Atra plus IDArubicin) trial for newly diagnosed APL. Results on over 800 patients showed a complete remission (CR) rate > 90% and an overall survival of 76% and confirmed that the concomitant administration of ATRA and chemotherapy is more effective than the sequential administration. Following the identification of distinct prognostic categories among APL patients, the GIMEMA group designed a new trial (AIDA2000) in which the intensity of post-remission treatment was adapted to the relapse risk and 498 patients were enrolled since January 2000. The results recently published showed a CR rate >90% with molecular remission rate after third consolidation of 98%. The new schedule allowed a Disease Free Survival (DFS) of 86% and showed that a risk-adapted strategy including ATRA for consolidation provides an outcome improvement in newly diagnosed patients. As reported by an international panel of experts, simultaneous ATRA and anthracycline chemotherapy schedules such as those used in the AIDA protocols represent the state of the art therapy for newly diagnosed APL.

ELIGIBILITY:
Inclusion Criteria:

* APL patients previously enrolled in the studies GIMEMA AIDA0493 and AIDA2000 surviving the initial diagnosis for more than 5 years and are in CR.
* Written informed consent provided.
* Adult patients at the time of registration onto this study.

Exclusion Criteria:

* Concomitant major psychiatric disorders or cognitive dysfunctions that would interfere with a self-reported evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute promyelocytic patients previously enrolled in the studies GIMEMA AIDA0493 and AIDA2000
Sampling Method: Non-Probability Sample
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Clinical significance on each of the SF-36 questionnaire scales. | One month from study entry.
  This will be performed by using HRQOL scores available for the Italian population. This will help identify which specific areas are mostly impaired and to what extent these patients recover in terms of HRQOL over the long run. This kind of comparison, which is only possible when HRQOL cultural-based norms are available, is largely used when investigating long-term HRQOL in cancer survivors and it is widely recognized as one of the most valuable approach in this kind of research setting.

SECONDARY OUTCOMES:
Association of EORTC-QLQC30 scales with social-demographic and clinical treatment related variables. | One month from study entry.
Association of MDASI scales (i.e., symptom severity and symptom interference) with different treatment strategies tested in the two GIMEMA trials. | One month from study entry.
Association of EORTC-QLQC30 scales with different treatment strategies tested in the two GIMEMA trials. | One month from study entry.
Association of rate of secondary malignancies with different treatment strategies tested in the two GIMEMA trials. | One month from study entry
Possible differences in EORTC-QLQC30, MDASI and SF-36 scales between patients who were less than eighteen years old at the time of diagnosis and patients who were at least eighteen years old at the time of diagnosis. | One month from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Principal Investigator — GIMEMA Foundation
Locations (38):
- Italy (38):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera - Nuovo Ospedale "Torrette", Ancona
  - Az.Ospedaliera S.G.Moscati, Avellino
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Divisione di Ematologia - Ospedali Riuniti, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria di Bolzano - Ospedale Centrale - Ematologia e Centro TMO, Bolzano
  - Spedali Civili - Brescia - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Policlinico di Careggi, Florence
  - Clinica Ematologica - DiMI - Università degli Studi di Genova, Genova
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - Divisione di Ematologia Ospedale "Santa Maria Goretti", Latina
  - Ospedale Niguarda " Ca Granda", Milan
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - N. Osp. divisione di Ematologia "S.Gerardo dei Tintori!", Monza
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Servizio Sanitario Nazionale - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" - Struttura Complessa di Ematologia - Div. TERE- 4° piano - Padiglione Palermo, Napoli
  - Sez. di Ematologia Clinica Ospedale San Francesco, Nuoro
  - Divisione di Ematologia con trapianto di midollo - A.U. Policlinico "Paolo Giaccone", Palermo
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Calabria Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - UOC Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, S. G. Rotondo
  - SCDO Ematologia 2 AOU S.Giovanni Battista, Torino
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza